CLINICAL TRIAL: NCT02502604
Title: Investigating the Efficacy of a Top-Down Approach to Cognitive Remediation in Individuals With Affective Disorders
Brief Title: Cognitive Training Program for Individuals With Depression and Post-Traumatic Stress Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Margaret McKinnon, Co-Chair, Research, Department of Psychiatry and Behavioural Neurosciences, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0416
Record Dates: First submitted 2015-07-15; First posted 2015-07-20 (Estimated); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Major Depressive Disorder; Post-traumatic Stress Disorder
Keywords: Cognitive Remediation; Goal Management Training; Major Depressive Disorder; Post-traumatic Stress Disorder; Neuropsychological Functioning
MeSH Terms: conditions — Depressive Disorder, Major; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Goal Management Training (Experimental): Participants in this arm of the study will attend GMT sessions, which will be administered weekly over a nine-week period following a script with accompanying slides and participant workbooks.
  Interventions: Behavioral: Goal Management Training
- Wait List Control (No Intervention): Participants in this category will be placed on a wait-list to receive goal management training following completion of their study participation.

INTERVENTIONS:
Behavioral: Goal Management Training — Goal management training sessions will be 2 hours in length and focus on learning skills that will assist in planning, carrying out, and monitoring goal-directed behaviours.
  Arms: Goal Management Training

SUMMARY:
Individuals with affective disorders (including post-traumatic stress disorder (PTSD) and major depressive disorder (MDD)) often experience declines in cognitive abilities such as memory and attention. Such difficulties can reduce functioning in important aspects of life, including at work or school. Little research has been conducted to investigate if cognitive dysfunction can be reduced in individuals with PTSD or MDD following a specific treatment. Thus, the investigators plan to determine the utility of a cognitive training program called goal management training (GMT) in reducing cognitive dysfunction in MDD/PTSD. GMT aims to assist participants in building skills in performing specific behaviours that rely on basic cognitive processes, allowing them to achieve an identified goal. 64 individuals with PTSD and 64 with MDD will be divided into two groups of 32, one GMT group, and one wait-list group that will receive GMT after study completion. The investigators predict that in comparison to the wait-list group, the GMT group will show greater improvements in cognitive functioning and everyday functioning following treatment and that these improvements will remain long-term.

DETAILED DESCRIPTION:
In addition to their core affective components, MDD and PTSD are associated with poor cognitive functioning across a host of highly similar domains, including declarative memory, short-term memory, attention, and executive functioning. These deficits have been associated with reduced response to pharmacological and non-pharmacological interventions and poor functional outcomes. Given the potentially devastating impact of poor cognitive functioning on the ability of patients with affective disorders to benefit from treatment interventions, and its association with poor functional outcomes, there is an urgent need to identify novel treatment interventions aimed at reducing cognitive dysfunction in these disorders. Accordingly, the aim of the present proposal is to a randomized controlled trial examining the efficacy of a well-established cognitive intervention aimed at reducing attentional and executive dysfunction, Goal Management Training® (GMT), in the treatment of cognitive deficits among patients with MDD and with PTSD. A secondary aim is to determine the longer-term impact of this approach on functional outcomes.

Importantly, limited investigation of cognitive remediation therapy has been performed in these populations. Only one study has been conducted to examine the impact of a non-standardized intervention protocol aimed at improving cognitive functioning in PTSD. Here, clinically (but not statistically) significant improvements were noted in a small pilot study on measures of cognitive functioning after employing bottom-up executive training approach in conjunction with transcranial direct current sample of four patients. Previously, the investigators have applied computer-assisted cognitive remediation, a bottom-up restitution based approach, in patients with MDD, resulting in improvements in performance on working memory tasks in conjunction with increased functional activity in lateral prefrontal and parietal areas, however, the broad benefits of this training observed in a small sample (n=12) did not generalize to a larger group.

GMT has demonstrated efficacy in several clinical and non-clinical populations that experience deficits in executive functioning, attention, and memory (similar to those seen in MDD and PTSD), including older adults, individuals who have suffered a traumatic brain injury, have attention-deficit hyperactivity disorder (ADHD), poly-substance abuse disorder, or spina bifida. In these studies, participants showed improvements in completing every-day tasks (as measured by self-report), as well as improvements in executive functions such as decision-making, working memory and selective attention. Critically, these results were maintained at follow-up (when assessed). Given the previous success of this intervention in remediating frontal-temporally mediated brain dysfunction across clinical populations, the investigators hypothesize that GMT has the ability to target similar cognitive difficulties experienced by those suffering from MDD and from PTSD. The investigators will further examine whether putative improvements in cognitive performance will translate to functional improvements analogous to those seen in other psychiatric populations undergoing cognitive remediation.

In the current study, the investigators will conduct the first study to investigate the utility of GMT in patients with MDD or with PTSD. Specifically, the primary aim of this proposed study is to examine whether a standardized 9-week program of GMT results in durable improvements in cognitive functioning relative to a wait-list control (WLC). A secondary aim will be to determine whether participation in the GMT group is associated with long-term functional improvements. The investigators hypothesize that at post-treatment, participants with MDD and with PTSD assigned to the GMT groups will show significantly greater improvement in neuropsychological test performance and greater functional improvement compared to participants in the WLC group; these gains are expected to be maintained at 3 month follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Structured Clinical Interview for DSM-IV-TR for Axis I Disorders (SCID-I (First et al., 1996))-confirmed primary diagnosis of MDD or PTSD
2. between the age of 18-60
3. able to provide written informed consent.

Exclusion Criteria:

1. Receiving treatment with anti-cholinergic or anti-psychotic medication
2. have had electroconvulsive therapy within the past year
3. a history of substance dependence or significant and recent (< 1 year) substance abuse)
4. a recent history (within the past 12 months) of medical disorder known to adversely affect cognition
5. loss of consciousness greater than 1 minute or a history of traumatic brain injury

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Verbal and Phonemic Fluency on the Controlled Oral Word Association Task | Change from baseline to 9 week and 3 month follow-ups.
Processing speed and response inhibition on the Stoop Colour and Word Test | Change from baseline to 9 week and 3 month follow-ups.
Attention alternation on the Trail Making Test Part B | Change from baseline to 9 week and 3 month follow-ups.
Forming and shifting concepts on the Wisconsin Card Sorting Task | Change from baseline to 9 week and 3 month follow-ups.
Processing speed on the Weschler Adult Intelligence Scale IV - Symbol Coding subtest | Change from baseline to 9 week and 3 month follow-ups.
Inattentiveness, impulsivity, sustained attention and vigilance on Connors Continuous Performance Task | Change from baseline to 9 week and 3 month follow-ups.
Working memory on the N-back Task | Change from baseline to 9 week and 3 month follow-ups.
  Measures ability to maintain and manipulate auditory information in memory.
Immediate and delayed memory, interference learning and recognition on the California Verbal Learning Test II | Change from baseline to 9 week and 3 month follow-ups.
Contextually based memory on the Weschler Memory Scale III - Logical Memory | Change from baseline to 9 week and 3 month follow-ups.
Nonverbal visuospatial memory on the Brief Visuospatial Memory Test - Revised | Change from baseline to 9 week and 3 month follow-ups.
Current intellectual functioning on the Weschler Abbreviated Scale of Intelligence - II | Baseline
Pre-morbid intellectual functioning on the National Adult Reading Test | Baseline
Self-reported executive difficulties on the Dysexecutive Questionnaire | Change from baseline to 9 week and 3 month follow-ups.
Self reported daily errors in distractibility, blunders, and memory on the Cognitive Failures Questionnaire | Change from baseline to 9 week and 3 month follow-ups.
Self reported work, education, and residential functioning on the Multidimensional Scale of Independent Functioning | Change from baseline to 9 week and 3 month follow-ups.
Disability in work, social relationships, and family life on the Sheehan Disability Scale | Change from baseline to 9 week and 3 month follow-ups.
Functional competence on the Canadian Objective Assessment of Life Skills - Brief Version | Change from baseline to 9 week and 3 month follow-ups.

SECONDARY OUTCOMES:
Current PTSD symptomatology on the Clinician Administered PTSD Scale for DSM 5 | Change from baseline to 9 week and 3 month follow-ups.
Exposure ot childhood trauma on the Childhood Trauma Questionnaire | Baseline
Dissociative symptoms on the Multiscale Dissociation Inventory | Change from baseline to 9 week and 3 month follow-ups.
Current depressive symptomatology on the Beck Depression Inventory - II | Change from baseline to 9 week and 3 month follow-ups.
Current anxiety symptomatology on the Beck Anxiety Inventory | Change from baseline to 9 week and 3 month follow-ups.

OTHER OUTCOMES:
Psychiatric diagnosis on the Structured Clinical Interview for DSM-IV - Text Revision | Baseline
  Assesses axis I disorders from the DSM-IV.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Jaeger J, Vieta E. Functional outcome and disability in bipolar disorders: ongoing research and future directions. Bipolar Disord. 2007 Feb-Mar;9(1-2):1-2. doi: 10.1111/j.1399-5618.2007.00441.x. No abstract available. PMID 17391343
- [Background] Marazziti D, Consoli G, Picchetti M, Carlini M, Faravelli L. Cognitive impairment in major depression. Eur J Pharmacol. 2010 Jan 10;626(1):83-6. doi: 10.1016/j.ejphar.2009.08.046. Epub 2009 Oct 14. PMID 19835870
- [Background] Polak AR, Witteveen AB, Reitsma JB, Olff M. The role of executive function in posttraumatic stress disorder: a systematic review. J Affect Disord. 2012 Dec 1;141(1):11-21. doi: 10.1016/j.jad.2012.01.001. Epub 2012 Feb 5. PMID 22310036
- [Background] Dunkin JJ, Leuchter AF, Cook IA, Kasl-Godley JE, Abrams M, Rosenberg-Thompson S. Executive dysfunction predicts nonresponse to fluoxetine in major depression. J Affect Disord. 2000 Oct;60(1):13-23. doi: 10.1016/s0165-0327(99)00157-3. PMID 10940443
- [Background] Altshuler LL, Bearden CE, Green MF, van Gorp W, Mintz J. A relationship between neurocognitive impairment and functional impairment in bipolar disorder: a pilot study. Psychiatry Res. 2008 Jan 15;157(1-3):289-93. doi: 10.1016/j.psychres.2007.01.001. Epub 2007 Sep 14. PMID 17868903
- [Background] Levine B, Stuss DT, Winocur G, Binns MA, Fahy L, Mandic M, Bridges K, Robertson IH. Cognitive rehabilitation in the elderly: effects on strategic behavior in relation to goal management. J Int Neuropsychol Soc. 2007 Jan;13(1):143-52. doi: 10.1017/S1355617707070178. PMID 17166313
- [Background] Levine B, Schweizer TA, O'Connor C, Turner G, Gillingham S, Stuss DT, Manly T, Robertson IH. Rehabilitation of executive functioning in patients with frontal lobe brain damage with goal management training. Front Hum Neurosci. 2011 Feb 17;5:9. doi: 10.3389/fnhum.2011.00009. eCollection 2011. PMID 21369362
- [Background] Levine B, Robertson IH, Clare L, Carter G, Hong J, Wilson BA, Duncan J, Stuss DT. Rehabilitation of executive functioning: an experimental-clinical validation of goal management training. J Int Neuropsychol Soc. 2000 Mar;6(3):299-312. doi: 10.1017/s1355617700633052. PMID 10824502
- [Background] Saunders N, Downham R, Turman B, Kropotov J, Clark R, Yumash R, Szatmary A. Working memory training with tDCS improves behavioral and neurophysiological symptoms in pilot group with post-traumatic stress disorder (PTSD) and with poor working memory. Neurocase. 2015;21(3):271-8. doi: 10.1080/13554794.2014.890727. Epub 2014 Feb 28. PMID 24579831
- [Background] Elgamal S, McKinnon MC, Ramakrishnan K, Joffe RT, MacQueen G. Successful computer-assisted cognitive remediation therapy in patients with unipolar depression: a proof of principle study. Psychol Med. 2007 Sep;37(9):1229-38. doi: 10.1017/S0033291707001110. Epub 2007 Jul 5. PMID 17610766
- [Background] Krasny-Pacini A, Limond J, Evans J, Hiebel J, Bendjelida K, Chevignard M. Context-sensitive goal management training for everyday executive dysfunction in children after severe traumatic brain injury. J Head Trauma Rehabil. 2014 Sep-Oct;29(5):E49-64. doi: 10.1097/HTR.0000000000000015. PMID 24495918
- [Background] In de Braek DMJM, Dijkstra JB, Ponds RW, Jolles J. Goal Management Training in Adults With ADHD: An Intervention Study. J Atten Disord. 2017 Nov;21(13):1130-1137. doi: 10.1177/1087054712468052. Epub 2012 Dec 20. PMID 23264370
- [Background] Stubberud J, Langenbahn D, Levine B, Stanghelle J, Schanke AK. Goal management training of executive functions in patients with spina bifida: a randomized controlled trial. J Int Neuropsychol Soc. 2013 Jul;19(6):672-85. doi: 10.1017/S1355617713000209. Epub 2013 Apr 11. PMID 23575309
- [Background] Alfonso JP, Caracuel A, Delgado-Pastor LC, Verdejo-Garcia A. Combined Goal Management Training and Mindfulness meditation improve executive functions and decision-making performance in abstinent polysubstance abusers. Drug Alcohol Depend. 2011 Aug 1;117(1):78-81. doi: 10.1016/j.drugalcdep.2010.12.025. Epub 2011 Feb 1. PMID 21277705
- [Derived] Cameron DH, McCabe RE, Rowa K, O'Connor C, McKinnon MC. A pilot study examining the use of Goal Management Training in individuals with obsessive-compulsive disorder. Pilot Feasibility Stud. 2020 Oct 6;6:151. doi: 10.1186/s40814-020-00684-0. eCollection 2020. PMID 33042571